CLINICAL TRIAL: NCT06575075
Title: A Double-blind, Placebo-controlled Study to Determine the Safety and Feasibility of Two Doses of Intravenous (2R, 6R)-Hydroxynorketamine (RR-HNK) in Adults With Obsessive-Compulsive Disorder
Brief Title: Pilot Study of RR-HNK in OCD
Acronym: (HNKO)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Carolyn Rodriguez (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Carolyn Rodriguez, Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 57628
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; AMPA receptor antagonist; hydroxynorketamine; ketamine metabolite
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — 6-hydroxynorketamine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized with a 1:1:1 allocation to either 0.25 mg/kg RR-HNK or 0.5 mg/kg IV RR-HNK + IV placebo (sterile saline)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.25 mg/kg RR-HNK (Experimental): OCD patients in this arm will receive 0.25mg/kg of RR-HNK - one single infusion. EEG and computerized behavioral tests will be acquired before and after infusion.
  Interventions: Drug: RR-HNK/Hydroxynorketamine
- 0.5 mg/kg RR-HNK (Experimental): OCD patients in this arm will receive 0.5mg/kg of RR-HNK - one single infusion. EEG and computerized behavioral tests will be acquired before and after infusion.
  Interventions: Drug: RR-HNK/Hydroxynorketamine
- Placebo (Sterile Saline) (Placebo Comparator): OCD patients in this arm will receive sterile saline - one single infusion. EEG and computerized behavioral tests will be acquired before and after infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RR-HNK/Hydroxynorketamine — (2R,6R)-Hydroxynorketamine is a metabolite of the drug ketamine and a glutamate AMPA receptor antagonist.
  Other Names: (2R,6R)-Hydroxynorketamine
  Arms: 0.25 mg/kg RR-HNK; 0.5 mg/kg RR-HNK
Drug: Placebo — Sterile Saline
  Arms: Placebo (Sterile Saline)

SUMMARY:
The purpose of this study is to understand how RR-HNK works in the brain to bring about a reduction in OCD symptoms.

DETAILED DESCRIPTION:
This protocol examines the safety and efficacy of 2 dosage levels of intravenous RR-HNK administration in individuals with OCD.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Meet the criteria for OCD diagnosis
* Failed at least 1 prior trial of standard first-line OCD treatment (e.g. SRI/CBT) or or had refused these treatments for individual reasons
* Agree to the following lifestyle modifications: comply with requirements for fasting prior to --the infusion session, not enroll in any other interventional clinical trials during the duration of the study, and commit to medication study procedures.
* Able to provide informed consent

Exclusion Criteria:

* Allergy or hypersensitivity to ketamine
* Any current or past medical/psychiatric condition that makes participation unsafe in the opinion of the investigator or study physician
* Pregnant or nursing, or able to become pregnant and are not practicing an effective means of birth control
* Lifetime history of deep brain stimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the severity of OCD symptoms as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS) | Baseline (Visit 3) to Week 1 (Visit 8), up to 1 week
  Change in OCD severity is measured by the YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response is defined as at least a 35% reduction on the YBOCS.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Rodriguez, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Phase 1 Assessment of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of (2R,6R)-Hydroxynorketamine in Healthy Volunteers — https://pubmed.ncbi.nlm.nih.gov/39054770/